CLINICAL TRIAL: NCT02390362
Title: Randomized Trial Comparing Rituximab Against Mycophenolate Mofetil in Children Wtih Refractory Nephrotic Syndrome (RAMP)
Brief Title: Randomized Trial Comparing Rituximab Against Mycophenolate Mofetil in Children Wtih Refractory Nephrotic Syndrome
Acronym: RAMP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding associated with enrollment milestones was withdrawn by Sponsor.
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Emory University (Other); Children's Healthcare of Atlanta (Other); Genentech, Inc. (Industry); The NephCure Foundation (Other)
Responsible Party: Principal Investigator, William Smoyer, William E. Smoyer, MD, Nationwide Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAMP001
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Frequent Relapsing Nephrotic Syndrome; Steroid Dependent Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Rituximab 375 mg/m2 will be administered intravenously on Study weeks 1 & 3.
  Interventions: Drug: Rituximab
- Mycophenolate Mofetil (MMF) (Active Comparator): Mycophenolate Mofetil will be continued in the patients in the MMF arm at a standard oral dose of 600 mg/m2 PO, BID starting on Study week 1 and continuing for 12 months
  Interventions: Drug: MMF

INTERVENTIONS:
Drug: Rituximab — We hypothesize that the anti-CD20 monoclonal antibody Rituximab will be more effective in maintaining remission in children who have already had one relapse while receiving MMF
  Arms: Rituximab
Drug: MMF — Subjects randomized to MMF, will continue MMF as scheduled by the investigator
  Arms: Mycophenolate Mofetil (MMF)

SUMMARY:
We hypothesize that the anti-CD20 monoclonal antibody Rituximab will be more effective than MMF in maintaining remission in children with frequent relapsing or steroid dependent nephrotic syndrome who have had one relapse while receiving MMF.

We will conduct a randomized study comparing two Rituximab infusions and continued MMF treatment. We plan to enroll 64 to have a comparater group of 58 (29 in each arm).

DETAILED DESCRIPTION:
After screening, and eligibility criteria have been met, children with steroid dependent and frequent relapsing nephrotic syndrome (SDNS and FRNS) will be enrolled into a 53 week study. The study is comprised of 3 sections; screening, treatment, and followup.

Screening will be <4 weeks from Day 1/week 1. Treatment is Day 1/Week 1 and Day 15/Week 3. Follow-Up is Week 7, Week 13, Week 19, Week 27 and Week 53. Participants will be randomized by the study pharmacy between screening and treatment Day1. If participant is randomized to Rituximab, then Treatment Day 15 will be based on tolerance of Rituximab infusion.

Safety assessments will occur at every visit beginning with Day 1.

ELIGIBILITY:
Inclusion Criteria:

* SDNS or FRNS
* Complete remission, defined by absence of edema and 3 consecutive daily urine dipstick readings of trace or negative for protein
* Must be taking MMF and have had at least one relapse while taking MMF in the prior 6 months that responded to corticosteroid treatment by re-entering complete remission at least 2 weeks prior to study entry.
* BMI prior to onset of NS <99th percentile
* Age 1-18 years
* Estimated GFR >40 ml/min/1.73m² (by Modified Schwartz formula)
* Negative serum pregnancy test (for females who are tanner stage 4 or 5)
* Males and females of reproductive potential (sexually active in boys or post-menarche in girls) must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment

Exclusion Criteria:

* • Prior therapy with rituximab, tacrolimus or cyclosporine

  * Prior therapy with cytotoxic agents in the past 90 days
  * History of genetic defects known to directly cause nephrotic syndrome (i.e. NPHS2 (podocin), NPHS1 (nephrin), PLCE1, WT1)
  * History of or concomitant severe, active infection (e.g. HIV, hepatitis B, hepatitis C)
  * History of diabetes mellitus
  * History of organ or bone marrow transplant
  * Secondary nephrotic syndrome (i.e. reflux nephropathy, IgA nephropathy, lupus nephritis, etc)
  * Live viral vaccines administered in the past 6 weeks (42 days)
  * Participation in another therapeutic trial within 30 days of enrollment
  * Allergy to study medications
  * ANC < 1.5 x 103
  * Hemoglobin: < 8.0 gm/dL
  * Platelets: < 100,000/mm
  * AST or ALT >2.5 x Upper Limit of Normal at the local institutions laboratory
  * Positive Hepatitis B or C serology (Hep B Surface antigen, Hep B Core antibody, and Hep C antibody)
  * History of HIV infection
  * Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
  * Receipt of a live vaccine within 4 weeks prior to randomization
  * Previous treatment with Natalizumab (Tysabri®)
  * Previous Treatment with Rituximab (Rituxan®)
  * Known hypersensitivity to Rituximab, to any of its excipients, or to murine proteins
  * History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
  * History of recurrent significant infection or history of recurrent bacterial infections
  * Known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
  * Lack of peripheral venous access
  * History of drug, alcohol, or chemical abuse within 6 months prior to screening
  * Pregnant, lactating, or refusal of birth control in an adolescent of child-bearing potential
  * Concomitant malignancies or previous malignancies
  * History of psychiatric disorder that would interfere with normal participation in this protocol
  * Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
  * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
  * Inability to comply with study and follow-up procedures

Patients who fail screening due to an abnormal laboratory parameter may be rescreened within the next 6 months if the local PI believes that the abnormality was transient and not related to a chronic underlying disease. Rescreening may only occur once and may not occur within 2 weeks of the initial screen failure.

If a patient has a clinically significant laboratory abnormality, the PI will be asked to define a follow-up plan (timing of repeating the laboratory test and/or additional work-up).

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12-07 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Smoyer, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital; Laurence Greenbaum, MD, Principal Investigator — University of Alberta
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only one site enrolled.
Period: Overall Study
Arm/Group | Rituximab | Mycophenolate Mofetil (MMF)
Started | 1 (1 subject enrolled in this arm. completed 2 doses of Rituximab.) | 2
Completed | 1 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Mycophenolate Mofetil (MMF) | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Relapse Free Survival
Time Frame: 6 months
Population: Study terminated early. Only three subjects were enrolled and results will not be posted to protect subject confidentiality.
Arm/Group | Rituximab | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Relapse Free at 12 Months
Time Frame: 12 months
Population: Study terminated early. Only 3 subjects enrolled. Data will not be posted to protect the subject identity.
Arm/Group | Rituximab | Mycophenolate Mofetil (MMF)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Rituximab | Mycophenolate Mofetil (MMF)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Study terminated early, sponsor pulled funding associated with enrollment milestones. At the time of termination, 2 subjects were active in the study. 1 was randomized to study drug, the other to the comparator drug. Not enough data for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes